CLINICAL TRIAL: NCT00569322
Title: Evaluation of Admission Blood Glucose Levels in the Intensive Care Unit
Brief Title: Admission Glucose ICU Study
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Other Study IDs: 01817-03-C
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2007-09

CONDITIONS: Hyperglycemia
Keywords: ICU; Admission; BG
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: BG Test

SUMMARY:
Determine if routine BG testing at the time of ICU admission is being done on all patients, irrespective of a prior diagnosis of diabetes mellitus, and whether it provides clinically important information.

DETAILED DESCRIPTION:
This prospective, observational study was performed in the medical-surgical ICU of a single hospital within a large multi-specialty healthcare system.

It was determined that it was not standard care to do glucose testing on all patients admitted to medical/surgical ICU's who did not have diagnosed diabetes and varied widely with the admitting service.

The primary objective of the study was to assess the availability and clinical value of blood glucose testing at the time of ICU admission after testing was implemented as routine care in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* ICU Admission

Exclusion Criteria:

* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2003-12; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa H Fish, MD, Principal Investigator — International Diabetes Center - Park Nicollet Health Services
Locations (1):
- Methodist Hospital - Park Nicollet Health Services, Minneapolis, Minnesota, United States